CLINICAL TRIAL: NCT05820659
Title: Racial Discrimination and Dysregulated Stress Response: Risk/Protective Factors
Brief Title: Racial Discrimination and Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U5GMACGETKJ1
Record Dates: First submitted 2023-03-29; First posted 2023-04-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-07

CONDITIONS: Stress Reaction; Acute
Keywords: cardiovascular reactivity; hypothalamic-pituitary-adrenal axis; inflammatory mediator; subtle racism
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stress inducing task (Experimental): Adolescents will complete an adapted peer rejection task on the computer to elicit the experience of subtle racial discrimination from White peers, as well as an impossible puzzle task to elicit cognitive stress.
  Interventions: Behavioral: peer rejection task and impossible puzzle task

INTERVENTIONS:
Behavioral: peer rejection task and impossible puzzle task — Peer rejection task: Adolescents will be informed that two peers will take turns to choose who they will chat with for different topics. Participants will not be chosen by virtual White peers 75% of the time. In reality, White peers are computerized avatars and whether or not adolescents are chosen by those peers is programmed with PsychoPy software.
  Impossible puzzle task: Adolescents will be asked to fit all puzzle pieces into a wooden frame with a wrong piece provided.

SUMMARY:
The goal of this study is to learn about whether ethnic minority adolescents' racial discrimination experience is related to dysregulated biological responses to subtle racism, and how the relationship may be attenuated or exacerbated by a set of social and cognitive factors. The main questions it aims to answer are:

* to reveal the relationship between racial discrimination experiences and ethnic minority adolescents' stress response to subtle racism
* to test parental ethnic-racial socialization, children's attribution to subtle racism and their racial identity as potential risk and protective factors.

DETAILED DESCRIPTION:
Racial discrimination experiences constitute significant risks for ethnic minority youth's physical and mental health problems. One explanation poses that chronic stress can lead to altered, dysregulated stress responses, which can make individuals susceptible to health problems. Currently, there is no experimental study that comprehensively measure ethnic minority youth's stress response to subtle racism, or investigate the contributing roles of racial discrimination experience and possible risk and protective factors.

A community sample of 9-14-year-old ethnic minority adolescents (40 Latino American, 40 Black/African American) and their parents will be recruited. The study employs an adapted peer rejection task which has been widely used with youth, and carefully designed to elicit the experience of subtle racial discrimination from White peers. Adolescents' cardiovascular activity and saliva samples will be taken at multiple time points before, during, and after the peer rejection task, tapping on response involving hypothalamic-pituitary-adrenal (HPA) axis, autonomic nervous system (ANS), and inflammatory mediator (IM). Adolescents will report their racial discrimination experience, make attribution about the peer rejection experience, report emotional experience, and rate their racial identity. Adolescents will complete an impossible puzzle task to elicit cognitive stress, during which they will be asked to fit all puzzle pieces into a wooden frame with a wrong piece provided. Their cardiovascular activity, attribution, and emotional experience in response to the impossible puzzle task will be measured. Parents will complete a questionnaire to report their ethnic-racial socialization practices.

The goals of this proposal are: 1) Reveal the relationship between racial discrimination experiences and ethnic minority adolescents' stress response to subtle racism as well as to cognitive stress; and 2) Test parental ethnic-racial socialization, children's attribution to subtle racism and their racial identity as potential risk and protective factors.

ELIGIBILITY:
Inclusion Criteria:

* 9-14 years old
* identified as Latino American or Black/African American
* Living in Warren county of Kentucky
* Parents of eligible adolescents

Exclusion Criteria:

Adolescents will not participate in the peer rejection task when they report to have:

* frequent experiences of peer victimization
* frequent experiences of racial discrimination
* severe depression
* severe social anxiety disorder
* severe generalized anxiety disorder

Ages: 9 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-11-17 (Actual)

PRIMARY OUTCOMES:
change in blood pressure for peer rejection | participants' blood pressure will be continuously monitored 5 minute before, during, and 45 minutes after the peer rejection task.
  participants' diastolic and systolic blood pressure will be continuously monitored.
change in stress hormones for peer rejection | participants' salivary samples will be collected at five time points (right before, 5 minutes after, 15 minutes after, 30 minutes after, and 45 minutes after the peer rejection task)
  participants' salivary samples will be collected, frozen, and assayed for cortisol.
change in inflammatory biomarker of Interleukin 6 for peer rejection | participants' salivary samples will be collected at five time points (right before, 5 minutes after, 15 minutes after, 30 minutes after, and 45 minutes after the peer rejection task)
  participants' salivary samples will be collected, frozen, and assayed for inflammatory biomarker of Interleukin-6
change in inflammatory biomarker of C-reactive protein for peer rejection | participants' salivary samples will be collected at five time points (right before, 5 minutes after, 15 minutes after, 30 minutes after, and 45 minutes after the peer rejection task)
  participants' salivary samples will be collected, frozen, and assayed for inflammatory biomarker of C-reactive protein
attribution about the peer rejection for peer rejection | right after the peer rejection task
  participants will complete the questionnaire, Attribution About The Peer Rejection (AATPR) to rate the likelihood of various reasons for the experience of peer rejection using a 7-point scale. The higher total score for the 4 racial reasons (possible range: 4-28) indicates the higher tendency of making racial attribution about the peer rejection.
emotional experience for peer rejection | right after the peer rejection task
  participants will complete the questionnaire, Emotions In The Peer Rejection (EITPR) to rate the emotional experiences in the peer rejection task using a 7-point scale. The higher total score for 5 sets of emotion terms (possible range: 5-35) indicates the higher levels of negative emotions in the peer rejection task.
change in skin conductance activity for peer rejection | participants' skin conductance will be continuously monitored 5 minutes before, during, and 45 minutes after the peer rejection task
  participants' skin conductance will be continuously monitored for the peer rejection task.
change in respiratory sinus arrhythmia for peer rejection | participants' electrocardiogram data will be continuously monitored 5 minutes before, during, and 45 minutes after the peer rejection task
  participants' electrocardiogram data that can be used to extract respiratory sinus arrhythmia, heart rate variability in synchrony with respiration, will be continuously monitored for the peer rejection task.

SECONDARY OUTCOMES:
change in cardiovascular activity for impossible puzzle | participants' systolic and diastolic blood pressure will be continuously monitored 5 minutes before, during, and 15 minutes after the impossible puzzle task
  participants' systolic and diastolic blood pressure will be continuously monitored for the impossible puzzle task
attribution for impossible puzzle | right after the impossible puzzle task
  participants will complete the questionnaire, Attribution About The Impossible Puzzle (AATIP) to rate the likelihood of various reasons for the experience of not being able to complete the puzzle using a 7-point scale. The higher total score for the 3 intrinsic reasons (possible range: 3-21) indicates the higher tendency of making intrinsic attribution about performance in the impossible puzzle task.
emotional experience for impossible puzzle | right after the impossible puzzle task
  participants will complete the questionnaire, Emotions In The Impossible Puzzle (EITIP) to rate the emotional experiences in the impossible puzzle task using a 7-point scale. The higher total score for 5 sets of emotion terms (possible range: 5-35) indicates the higher levels of negative emotions in the impossible puzzle task
change in skin conductance for impossible puzzle | participants' skin conductance will be continuously monitored 6 minutes before, during, and 15 minutes after the impossible puzzle task
  participants' skin conductance will be continuously monitored for the impossible puzzle task
change in respiratory sinus arrhythmia for impossible puzzle | participants' electrocardiogram data will be continuously monitored 6 minutes before, during, and 15 minutes after the impossible puzzle task
  participants' electrocardiogram data that can be used to extract respiratory sinus arrhythmia, heart rate variability in synchrony with respiration, will be continuously monitored for the impossible puzzle task

CONTACTS AND LOCATIONS:
Overall Officials: Qingfang Song, Ph.D, Principal Investigator — Western Kentucky University
Locations (1):
- Western Kentucky University, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The research resources from the project will include the study protocol and associated data, which will be provided upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The protocol and deidentified data will become available six months after the first publication.
Access Criteria: Data will be shared upon individual request.

REFERENCES:
- [Background] Lucas T, Wegner R, Pierce J, Lumley MA, Laurent HK, Granger DA. Perceived Discrimination, Racial Identity, and Multisystem Stress Response to Social Evaluative Threat Among African American Men and Women. Psychosom Med. 2017 Apr;79(3):293-305. doi: 10.1097/PSY.0000000000000406. PMID 27806018
- [Background] Silk JS, Stroud LR, Siegle GJ, Dahl RE, Lee KH, Nelson EE. Peer acceptance and rejection through the eyes of youth: pupillary, eyetracking and ecological data from the Chatroom Interact task. Soc Cogn Affect Neurosci. 2012 Jan;7(1):93-105. doi: 10.1093/scan/nsr044. Epub 2011 Jul 20. PMID 21775386
- [Background] Sladek MR, Castro SA, Doane LD. Ethnic-Racial discrimination experiences predict Latinx adolescents' physiological stress processes across college transition. Psychoneuroendocrinology. 2021 Jun;128:105212. doi: 10.1016/j.psyneuen.2021.105212. Epub 2021 Apr 1. PMID 33933893